CLINICAL TRIAL: NCT01771289
Title: Phase II Trial of Neoadjuvant Concurrent Chemoradiation With Weekly Docetaxel/Cisplatin for Resectable IIIA-N2 NSCLC
Brief Title: Neoadjuvant Concurrent Chemoradiation With Weekly Docetaxel/Cisplatin for Resectable IIIA-N2 NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Principal Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-XW1301
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemoradiation (Experimental)
  Interventions: Drug: docetaxel/cisplatin; Radiation: Radiation

INTERVENTIONS:
Drug: docetaxel/cisplatin — weekly docetaxel/cisplatin combined with radiation
Radiation: Radiation — chemoradiation

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of neoadjuvant concurrent chemoradiation with weekly docetaxel/cisplatin in patients with resectable IIIA-N2 NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years older.
* Present with histologically proven or cytological diagnosis of NSCLC Stage IIIA as defined by the American Joint Committee on Cancer Staging Criteria for Lung Cancer, that is amenable to surgery.
* No prior systemic chemotherapy or targeted therapy for lung cancer before screening.
* ECOG performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* Adequate hematological function:Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).
* Adequate liver function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN);Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in subjects without liver metastases; ≤ 5 x ULN in subjects with liver metastases.
* Adequate renal function:Serum creatinine ≤ 1.25 x ULN, and creatinine clearance ≥ 60 ml/min.
* Female subjects should not be pregnant or breast-feeding.

Exclusion Criteria:

* Patients with prior exposure to agents directed at the HER axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior chemotherapy or therapy with systemic anti-tumour therapy (e.g. monoclonal antibody therapy).
* History of another malignancy in the last 5 years with the exception of the following:Other malignancies cured by surgery alone and having a continuous disease-free interval of 5 years are permitted; Cured basal cell carcinoma of the skin and cured in situ carcinoma of the uterine cervix are permitted.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Known hypersensitivity to Tarceva or gemcitabine or cisplatin.
* Eye inflammation or eye infection not fully treated or conditions predisposing the subject to this.
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicated the use of an investigational drug or puts the subject at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
downstage rate of mediastinal lymph nodes | 8 weeks

SECONDARY OUTCOMES:
overall survival | 5y
Disease-free survival | 5y
resection rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China